CLINICAL TRIAL: NCT03074552
Title: Probiotic Prophylaxis for Microbiome Modulation and Ventilator Associated Pneumonia (VAP) or Severe Infections Prevention in Multitrauma Patients: a Multicenter, Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Probiotic Prophylaxis for Microbiome Modulation and VAP or Infections Prevention in Multitrauma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Uni-Pharma (Industry)
Responsible Party: Principal Investigator, Georgia Tsaousi, Assistant Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ProVAP
Record Dates: First submitted 2017-02-25; First posted 2017-03-09 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Ventilator Associated Pneumonia; Infection; Trauma
Keywords: probiotics; VAP; microbiome; trauma; infections
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Infections; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The present study will be a multicenter, randomized, double-blind, placebo-controlled trial including data collected from 9 ICUs. Patients will be randomly assigned in a 1:1 ratio to receive probiotic or placebo treatment according to a computer-based table blinded to study investigators and physicians in charge.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A numbered sealed envelope will be used to ensure blinding. Only the pharmacist responsible for the sealed envelopes preparation will be aware of its content, with no further involvement in the study protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): The probiotic preparation [ LactoLevure] will consist a combination of four probiotics.
  Interventions: Dietary Supplement: LactoLevure
- Placebo (Placebo Comparator): Placebo will consist of identical capsules of powdered glucose polymer, and they will be constructed by the same industry that manufactures the probiotics capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: LactoLevure — The probiotic preparation will consist a combination of four probiotics: Lactobacillus acidophilus LA-5 1.75 × 109 CFU, Lactobacillus Plantarum 0.5 × 109 CFU, Bifidobacterium lactis BB-12 1.75 × 109 CFU και Saccharomyces boulardii 1.5 × 109 CFU per capsule (LactoLevure, UniPharma, Athens, Greece).
  Arms: Probiotics
Other: Placebo — Placebo will consist of identical capsules of powdered glucose polymer
  Arms: Placebo

SUMMARY:
Ventilator-associated pneumonia (VAP), is a type of pneumonia that develops more than 48 hours after endotracheal intubation, is common in intensive care units (ICUs). It is estimated to be responsible for 27% to 47% of ICU-acquired infections.

The pathogenesis of VAP is complex but typically involves colonization of the aerodigestive tract with pathogenic bacteria, the formation of biofilms, and microaspiration of contaminated secretions. Preventing carriage of potentially pathogenic micro-organisms from the aerodigestive tract is an infection control strategy used to reduce the occurrence of VAP. One novel intervention is the administration of prophylactic probiotics which restore non-pathogenic flora that compete with pathogens, modulate local and systemic immunity, and decrease intestinal permeability and thus can be beneficial in preventing nosocomial infections in critically ill patients. The role of the probiotics in preventing VAP in mechanically ventilated patients is inconclusive. Some evidence indicates that probiotics may reduce the incidence of VAP by inhibiting pathogen adhesion, improving gut mucosal barrier function, reducing bacterial translocation and up-regulating the immune system. Furthermore, guidelines remain inconclusive regarding the role of commensal oropharyngeal flora (COF) as a causative agent in VAP, mainly due to a scarcity of studies in this research field. However, there is evidence that COF may cause pulmonary infection, mostly in immunocompromised patients.

DETAILED DESCRIPTION:
The oropharyngeal swab will be collected on days 1, 3 and 7 after ICU admission and upon the occurrence of VAP or other infection. Nonbronchoscopic bronchoalveolar lavage (BAL) using a protected catheter will be collected on day 3 after ICU admission and upon the occurrence of VAP. Whole blood sample and stool sample will be collected on day 1 after ICU admission and upon the occurrence of VAP or other infection for microbiome analysis.

As soon as the first sample of the oropharyngeal swab is collected, patients will be allocated to the "treatment" groups. Each patient will receive two capsules per day for 15 consecutive days post admission. The content of one capsule will be suspended in 100ml tap water and administered by nasogastric tube or through), while the content of the other capsule will be suspended in sterile, water-based surgical lubricant and administered as a slurry to the oropharynx. The administration will be performed by a study nurse who was responsible for ascertaining that the whole prepared volume is given.

The study protocol-mandated baseline data will include demographic information, medical history, and the APACHE II, SAPS II, NISS and SOFA score, and Operative POSSUM score (only cases undergoing surgical treatment).

Additional information collected on a daily basis will include patient's clinical course with special emphasis on clinical signs of VAP or infections, type of chemoprophylaxis, endotracheal or tracheostomy tube cuff pressure, type of nutrition and bowel movement. Furthermore, duration of intubation, tracheostomy day after ICU admission, duration of mechanical ventilation, lengths of stay in the ICU and hospital, adverse events (related and non-related to probiotics administration) and mortality. Data recording will be extended up to 30 days after hospital admission (patient recovered, treated in ICU / department or death).

Central venous line infection will be considered as positive when there is bacteremia with common skin commensal and positive catheter tip culture or exit site culture for the same organism.

An ICU-acquired urinary tract infection will be deemed present if there are at least 103 colony-forming units (cfu)/mL of 1 or 2 micro-organisms identified by urine culture in patients who develop a positive urine culture first identified 48 h or later after ICU admission.

A superficial incisional infection (SSI) must meet the following criterion:

Infection occurs within 30 days after the operative procedure and involves only skin and subcutaneous tissue of the incision and patient has at least 1 of the following:

* purulent drainage from the superficial incision
* organisms isolated from an aseptically obtained culture of fluid or tissue from the superficial incision
* at least 1 of the following signs or symptoms of infection: pain or tenderness, localized swelling, redness, or heat, and superficial incision is deliberately opened by the surgeon and is culture positive or not cultured. A culture-negative finding does not meet this criterion.
* diagnosis of superficial incisional SSI by the surgeon or attending physician.

Intraabdominal trauma infection will be defined by the following:

* Temperature >38°C or <36°C
* White blood cell count >12 000/mm3 or <4000/mm3 or >10% immature bands
* Abdominal tenderness during clinical examination
* CT scanning compatible with positive findings for acute intraabdominal infection An antibiotics-related infection will be documented by the detection of toxins produced by C. difficile bacteria in a stool sample.

Bacteremia will be defined as the presence of a recognized Gram(+) or Gram(-) pathogen or Candida spp cultured from one or more blood cultures and organism cultured from blood is not related to an infection at another site Sepsis is defined as life-threatening organ dysfunction caused by a dysregulated host response to infection.

Organ dysfunction will be identified as an acute change in total SOFA score ≥2 points consequent to the infection.

Patients with septic shock will be identified with a clinical construct of sepsis with persisting hypotension requiring vasopressors to maintain MAP ≥65 mm Hg and having a serum lactate level >2 mmol/L (18mg/dL) despite adequate volume resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* adults >18 and < 80 years oldmultitrauma patients with at least two organ-system injury
* intubated immediately after injury
* likelihood that the patient would require mechanical ventilation with an endotracheal tube (or tracheostomy) for >10 days
* life expectancy > 15 days

Exclusion Criteria:

* investigators unable to obtain informed written consent from patients' relatives
* administer the first dose of the study drug within 24 hours of intubation
* pregnancy; lactation; immunosuppression; hematologic disease; prosthetic cardiac valve or vascular graft; cardiac trauma; history of rheumatic fever, endocarditis, or congenital cardiac abnormality; oropharyngeal mucosal injury; recent history of sinusitis and respiratory tract infection
* obesity [BMI > 40]
* administration of antibiotics for > 3 days before recruitment into the study
* administration of probiotics before recruitment into the study
* history of infection from Hepatis B or C and HIV
* administration of < 90% of the predicted doses of probiotics during the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-08-19 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Probiotics for VAP prophylaxis | 30 days
  To determine the efficacy of probiotic administration for the prophylaxis of VAP in a multi trauma population admitted in the ICU This outcome will be assessed by the difference of number of cases (n) and percentage of change (%) in VAP development between probiotics and control groups
  Ventilator associated pneumonia (VAP) will be defined as pneumonia developing more than 48 h after endotracheal intubation and initiation of mechanical ventilation. The diagnostic criteria for VAP will be the following:
  * SOFA score elevation of at least 1 point
  * New or progressive radiographic consolidation or infiltrate. In addition, at least 2 of the following:
    * Temperature > 38 °C
    * Leukocytosis (white blood cell count ≥ 12,000 cells/ mm3) or leukopenia (white blood cell count < 4,000 cells/mm3)
    * Presence of purulent secretions
  * BAL > 104 colony forming units (CFU)/ml)

SECONDARY OUTCOMES:
Probiotics for indections control | 30 days
  The efficacy of probiotics for controlling infections related to trauma, urinary tract, central venous line or related to antibiotics use.
  This outcome will be assessed by the difference of number of cases (n) and percentage of change (%) in infections other than VAP between probiotics and control groups [The criteria for documentation of the above-mentioned infections are provided in more detail in the Detailed Description section]
Probiotics for bacteremia, sepsis or septic shock reduction | 30 days
  The efficacy of the use of probiotics for reducing the incidence of bacteremia, sepsis or septic shock.
  This outcome will be assessed by the difference of number of cases (n) and percentage of change (%) in bacteremia, sepsis or septic shock between probiotics and control groups [The criteria for documentation of the above-mentioned infections are provided in more detail in the Detailed Description section].

OTHER OUTCOMES:
Impact of Probiotics use on parameters related to hospitalization and mortality | 30 days
  The difference of duration of mechanical ventilation (days), the length of ICU stay (days) and of total hospitalization (days), between probiotics and control group will be assessed. Moreover, the difference of the number (n) and percentage (%) of the deaths recorded between probiotics and control group up to 30 days after ICU admission.

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Kotzampassi, MD, PhD, Study Director — Aristotle University Of Thessaloniki
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scholte JB, van der Velde JI, Linssen CF, van Dessel HA, Bergmans DC, Savelkoul PH, Roekaerts PM, van Mook WN. Ventilator-associated Pneumonia caused by commensal oropharyngeal Flora; [corrected] a retrospective Analysis of a prospectively collected Database. BMC Pulm Med. 2015 Aug 12;15:86. doi: 10.1186/s12890-015-0087-y. PMID 26264828
- [Background] Wang J, Liu KX, Ariani F, Tao LL, Zhang J, Qu JM. Probiotics for preventing ventilator-associated pneumonia: a systematic review and meta-analysis of high-quality randomized controlled trials. PLoS One. 2013 Dec 18;8(12):e83934. doi: 10.1371/journal.pone.0083934. eCollection 2013. PMID 24367620
- [Background] Zeng J, Wang CT, Zhang FS, Qi F, Wang SF, Ma S, Wu TJ, Tian H, Tian ZT, Zhang SL, Qu Y, Liu LY, Li YZ, Cui S, Zhao HL, Du QS, Ma Z, Li CH, Li Y, Si M, Chu YF, Meng M, Ren HS, Zhang JC, Jiang JJ, Ding M, Wang YP. Effect of probiotics on the incidence of ventilator-associated pneumonia in critically ill patients: a randomized controlled multicenter trial. Intensive Care Med. 2016 Jun;42(6):1018-28. doi: 10.1007/s00134-016-4303-x. Epub 2016 Apr 4. PMID 27043237
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Shankar-Hari M, Phillips GS, Levy ML, Seymour CW, Liu VX, Deutschman CS, Angus DC, Rubenfeld GD, Singer M; Sepsis Definitions Task Force. Developing a New Definition and Assessing New Clinical Criteria for Septic Shock: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):775-87. doi: 10.1001/jama.2016.0289. PMID 26903336
- [Background] Kotzampassi K, Giamarellos-Bourboulis EJ. Probiotics for infectious diseases: more drugs, less dietary supplementation. Int J Antimicrob Agents. 2012 Oct;40(4):288-96. doi: 10.1016/j.ijantimicag.2012.06.006. Epub 2012 Aug 2. PMID 22858373
- [Background] Stavrou G, Giamarellos-Bourboulis EJ, Kotzampassi K. The role of probiotics in the prevention of severe infections following abdominal surgery. Int J Antimicrob Agents. 2015 Dec;46 Suppl 1:S2-4. doi: 10.1016/j.ijantimicag.2015.10.003. PMID 26686273
- [Background] Kotzampassi K, Stavrou G, Damoraki G, Georgitsi M, Basdanis G, Tsaousi G, Giamarellos-Bourboulis EJ. A Four-Probiotics Regimen Reduces Postoperative Complications After Colorectal Surgery: A Randomized, Double-Blind, Placebo-Controlled Study. World J Surg. 2015 Nov;39(11):2776-83. doi: 10.1007/s00268-015-3071-z. PMID 25894405
- [Background] Giamarellos-Bourboulis EJ, Bengmark S, Kanellakopoulou K, Kotzampassi K. Pro- and synbiotics to control inflammation and infection in patients with multiple injuries. J Trauma. 2009 Oct;67(4):815-21. doi: 10.1097/TA.0b013e31819d979e. PMID 19820590